CLINICAL TRIAL: NCT05516797
Title: Continuous Glucose Monitoring Versus Blood Glucose Monitoring to Optimize Glycemic Outcomes in People With Type 2 Diabetes Following the Virta Treatment Program" (IGNITE: Impact of Glucose moNitoring and nutrItion on Time in rangE Study)
Brief Title: IGNITE (Impact of Glucose moNitoring and nutrItion on Time in rangE)
Acronym: IGNITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Virta Health (Industry); Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A22-076
Record Dates: First submitted 2022-08-09; First posted 2022-08-26 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: Continuous Glucose Monitoring (CGM); Blood Glucose Monitoring (BGM); Nutrition Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Continuous Glucose Monitoring (CGM) (Experimental): Participants in this arm will use the FreeStyle Libre 2 CGM sensor.
  Interventions: Device: Continuous Glucose Monitoring (CGM)
- Blood Glucose Monitoring (BGM) (No Intervention): Participants in this arm will use the Precision Xtra fingerstick blood glucose meter throughout the study.

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — Use of CGM (FreeStyle Libre 2) compared to BGM for glucose monitoring
  Arms: Continuous Glucose Monitoring (CGM)

SUMMARY:
The purpose of this study is to learn whether there is a difference in the amount of time glucose (blood sugar) stays within a target range (glucose 70 - 180 mg/dl) when using either continuous glucose monitoring (CGM) or fingerstick blood glucose monitoring (BGM) in people with Type 2 diabetes who participate in the Virta Treatment program.

DETAILED DESCRIPTION:
The purpose of this three-month, randomized, controlled trial is to compare the difference in change in 14-day CGM-derived TIR (% time with glucose 70-180 mg/dL) from Baseline to 3-months Post-Dietary Change in participants with T2D who are assigned to use either BGM or CGM. The difference in mean blood ketone levels and additional glycemic endpoints will also be compared, and several exploratory endpoints, including medication changes, dietary intake, and body weight will be described.

The study also includes a three-month Follow-Up period (months three to six), where participants will remain using their randomly assigned glucose monitoring modality (e.g., BGM or CGM); this period will help assess durability of the results found during the intervention.

This study will provide insights into how continuous feedback from CGM affects glycemic outcomes, such as TIR and HbA1c, compared to the standard method of BGM. It is important to understand if the methods of glucose monitoring differ, because greater TIR and lower HbA1c are associated with reduced risk of diabetes complications.

While many studies have compared the differences in glycemic outcomes between BGM and CGM, this study compares differences between the two glucose monitoring methods as part of a randomized, controlled intervention in people with T2D where dietary patterns will be adjusted. It is possible that this study will help demonstrate whether the continuous feedback provided by CGM influences adherence to dietary guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. U.S. residence with plans to remain in the U.S. for study duration (for shipping purposes)
3. Diagnosis of T2D
4. HbA1c between 7.5-11.5% documented within 60 days prior to consent
5. Stable diabetes medication regimen and lifestyle patterns (eating and activity) within approximately 90 days prior to consent
6. Using at least one glucose-lowering medication (oral or injectable) for diabetes management at the time of consent; if using insulin, this may include up to a total of three or fewer insulin injections per day (e.g., once or twice daily basal insulin, once or twice daily basal insulin plus one prandial insulin dose, once or twice daily pre-mix insulin, or another combination etc.)
7. English language comprehension
8. Confirmed download of FreeStyle Libre 2 app on personal smartphone with access to WiFi
9. Willing and able to record study data using smartphone, tablet, and/or computer
10. Willing to wear and use study-provided CGM devices for up to 7 months
11. Willing to perform fingersticks to test blood glucose
12. Willing to perform fingersticks to test blood ketones twice daily
13. Eligible to initiate and intention to participate in the dietary changes required as part of the Virta Treatment for at least 7 months

Exclusion Criteria:

1. Type 1 diabetes
2. Currently using an insulin pump or multiple daily injection insulin therapy with >3 insulin injections per day or using bolus injections to cover every meal
3. Currently following a self-reported, very low-carbohydrate eating pattern
4. Currently using a personal CGM or plans to use a personal CGM during the study period
5. Advanced-stage renal, cardiac, hepatic, or other chronic disease
6. History of ketoacidosis
7. Pregnant, lactating, or planned pregnancy
8. Allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin
9. Participation in another interventional trial at the time of enrollment or during the study period
10. Participant is unsuitable for participation due to any cause as determined by Investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Willis, PhD, Principal Investigator — HealthPartners Institute dba International Diabetes Center
Locations (1):
- Health Partners Institute dba International Diabetes Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were required to complete a baseline assessment period prior to beginning the intervention. This included wearing a blinded CGM for up to 14-days along with assessment of HbA1c and completion of several surveys. More participants were enrolled than were randomized. Some participants who enrolled did not complete the required baseline assessment requirements for randomization or they voluntarily withdrew before randomization. This is why N=178 enrolled and N=163 were randomized.
Groups:
- Continuous Glucose Monitoring (CGM) Arm: Participants in this arm took part in a medically supervised ketogenic diet program. They wore and used a Freestyle Libre 2 continuous glucose monitoring system on thier personal smartphone during the entire intervention period.
- Blood Glucose Monitoring (BGM) Arm: Participants in this arm took part in a medically supervised ketogenic diet program. The BGM arm participants used a Precision Xtra Blood Glucose and Ketone Monitoring System (Abbott Diabetes Care) daily; fingerstick glucose testing was prescribed on an individual basis. Participants in this arm also wore a blinded Freestyle Libre Pro continuous glucose monitoring system during specified intervals throughout the intervention period.
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Started | 81 | 82
Completed | 72 | 64
Not Completed | 9 | 18

BASELINE CHARACTERISTICS:
Population: Information about the analyzed population matches the number of participants assigned to each arm. Analysis information is presented for N=81 in CGM and N=82 in BGM.
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm | Total
Number analyzed (Participants) | 81 | 82 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.7) | 52.3 (9.3) | 52.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 40 | 44 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 9 | 13 | 22
  White | 62 | 59 | 121
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 3 | 6
Hb1ac [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 8.1 (1.2) | 8.1 (1.2) | 8.1 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Change in 14-day CGM-derived TIR From (3 Months Minus Baseline)
Description: Change in 14-day CGM-derived TIR (% time with glucose 70-180 mg/dL) from Baseline to 3-month Post-Dietary Change period between participants with T2D who are randomized to use either BGM or CGM (3 months minus baseline)
Time Frame: Three (3) months
Population: Participants with adequate blinded CGM data at baseline and at month 3 were included.
Measure: Mean (95% Confidence Interval); unit: percentage of time with glucose 70-180 m
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 72 | 64
percentage of time with glucose 70-180 m | 28 [21 to 34] | 22 [15 to 29]

2. Secondary Outcome: 90-day Mean Blood Ketone Levels
Description: Mean of blood ketone levels from day 0 to day 90 (three months).
Time Frame: Three (3) months / 90 days
Population: Results from general and generalized linear mixed models using all available data
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 79 | 81
mmol/L | 0.54 [0.47 to 0.61] | 0.48 [0.42 to 0.55]

3. Secondary Outcome: Participants Reaching CGM-derived Consensus Targets
Description: Percent of participants reaching CGM-derived consensus targets (targets defined as meeting both >70% TIR70-180 mg/dL and <4% TBR <70mg/dL) at the end of the 3-month Post-Dietary in both the BGM and CGM arms
Time Frame: Three (3) months
Population: Some data missing at random; used all available and qualifying data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 72 | 64
percentage of participants | 81 [70 to 89] | 66 [53 to 78]

4. Secondary Outcome: Difference in Change in HbA1c
Description: Change in HbA1c from Baseline to the end of the 3-month Post-Dietary Change period between BGM and CGM arms
Time Frame: Three (3) months
Population: Some data missing at random; all available and qualifying data were used
Measure: Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 64 | 64
percentage of glycated hemoglobin | -1.6 [-1.8 to -1.3] | -1.5 [-1.7 to -1.2]

5. Other Pre Specified Outcome: Difference in Change in CGM-derived Metric %Time Above Range >180 mg/dL During 3-month Post-Dietary Change Period (3 Month Minus Baseline)
Description: Change in the % time above range >180 mg/dL, during the Baseline to 3-month Post-Dietary Change period for both arms (3 months minus baseline)
Time Frame: Three (3) months
Population: Some data were missing at random; analysis used all available qualifying data
Measure: Mean (95% Confidence Interval); unit: percent time with glucose >180mg/dL
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 72 | 64
percent time with glucose >180mg/dL | -28 [-34 to -21] | -23 [-30 to -17]

6. Other Pre Specified Outcome: Difference in Change in the CGM-derived Metric, %Time Below Range <70 mg/dL (3 Months Minus Baseline)
Description: Change in %Time below range <70 mg/dL during the Baseline to 3-month Post-Dietary Change period (3 months minus baseline)
Time Frame: 3 months (baseline to three months)
Population: some data missing at random; all available and qualifying data were used
Measure: Mean (95% Confidence Interval); unit: percent time with glucose <70mg/dL
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 72 | 64
percent time with glucose <70mg/dL | 0.7 [0 to 1.5] | 1.2 [0.4 to 2.0]

7. Other Pre Specified Outcome: Difference in Change in the CGM-derived Metric %Time Below Range <54 mg/dL, From Baseline to 3-month Post-Dietary Change Period (3 Months Minus Baseline)
Description: Change in % Time with glucose below range <54 mg/dL from Baseline to 3-month Post-Dietary Change (3 months minus baseline)
Time Frame: Three (3) months (baseline to three months)
Population: some data missing at random; all available and qualifying data were used
Measure: Mean (95% Confidence Interval); unit: percent time with glucose <54 mg/dL
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 72 | 64
percent time with glucose <54 mg/dL | -0.01 [-0.09 to 0.06] | 0.04 [-0.09 to 0.06]

8. Other Pre Specified Outcome: Difference in Change in the CGM-derived Metric, Mean Sensor Glucose, From Baseline to 3-month Post-Dietary Change Period (3 Months Minus Baseline)
Description: Change in the CGM-derived metric, Mean sensor glucose, from baseline to three months
Time Frame: Three (3) months (baseline to three months)
Population: some data missing at random; all available and qualifying data were used
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 72 | 64
mg/dL | -48 [-58 to -37] | -42 [-53 to -31]

9. Other Pre Specified Outcome: Difference in Change in the CGM-derived Metric, % Coefficient of Variation, From Baseline to 3-month Post-Dietary Change Period (3 Months Minus Baseline)
Description: Change in % Coefficient of variation from Baseline to 3-month Post-Dietary Change (3 months minus baseline)
Time Frame: Three (3) months (baseline to three months)
Population: some data missing at random; all available and qualifying data were used
Measure: Mean (95% Confidence Interval); unit: percent of coefficient of variation
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
Number analyzed (Participants) | 72 | 64
percent of coefficient of variation | -4 [-6 to -3] | -4 [-5 to -2]

ADVERSE EVENTS:
Time Frame: Adverse and Serious adverse events were collected from the time of consent through the end of study completion, this is approximately seven months for each participant when considering the baseline assessment period and the intervention period.
Description: AEs were defined as (1) severe CGM sensor-related reactions/infections requiring in-person medical care, (2) severe hypoglycemia that required assistance of another person due to altered consciousness or (3) severe hyperglycemia if the event involved diabetic ketoacidosis hyperosmolar or hyperglycemic state, as defined by Kitabchi et al. SAEs were defined as anything serious, unexpected, and probably, possibly, or definitely related to the glucose monitoring device or research procedures.
Arm/Group | Continuous Glucose Monitoring (CGM) Arm | Blood Glucose Monitoring (BGM) Arm
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/82
Other Adverse Events (participants affected / at risk) | 0/81 | 0/82

LIMITATIONS AND CAVEATS:
CGM was compared with BGM in people with T2D; however, many people with T2D do not regularly use glucose monitoring, it would have been ideal to compare both groups to a third arm that was not using any glucose monitoring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT05516797/Prot_SAP_001.pdf